CLINICAL TRIAL: NCT06553768
Title: Randomized Double-Blind Placebo-Controlled Phase 3 Study to Evaluate the Efficacy and Safety of Maralixibat in the Treatment of Participants With Cholestatic Pruritus
Brief Title: Evaluation of Maralixibat in Pruritus Associated With General Cholestatic Liver Disease (EXPAND)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Mirum Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MRX-802; 2024-511287-85-00 (EU CTIS Number)
Record Dates: First submitted 2024-08-08; First posted 2024-08-14 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Cholestatic Liver Disease (Except ALGS, PFIC, PBC and PSC)
Keywords: Pruritus; Cholestatic Liver Disease; Biliary Atresia
MeSH Terms: conditions — Cholangitis, Sclerosing; Pruritus; Biliary Atresia | interventions — maralixibat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Maralixibat (Experimental): Participants will receive maralixibat oral solution 300 μg/kg orally once daily for 1 week and then twice daily for 39 weeks.
  Interventions: Drug: Maralixibat
- Placebo (Placebo Comparator): Participants will receive placebo matched to maralixibat oral solution orally once daily for 1 week and then twice daily for 19 weeks. After 20 weeks, participants will receive maralixibat oral solution 300 μg/kg orally once daily for 1 week and then twice daily for 19 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Maralixibat — Maralixibat will be provided as an oral solution along with 0.5-, 1.0-, and 3.0-mL sized dosing dispensers. During the double-blind dose escalation period (4 weeks), the study drug (maralixibat) will be administered once daily for 1 week and then twice daily (BID; morning and evening). During the double-blind stable dosing period (16 weeks), participants will be treated with 300 μg/kg BID or the maximum tolerated dose (determined during the double-blind dose-escalation period) of maralixibat. During the open-label dose escalation period (4 weeks), all participants will receive maralixibat treatment once daily for 1 week and then twice daily (BID; morning and evening). During the open-label stable dosing period (at least 16 weeks), participants will be treated with 300 μg/kg BID or the maximum tolerated dose (determined during the open-label dose-escalation period) of maralixibat.
  Other Names: Formerly LUM001, SHP625
  Arms: Maralixibat
Other: Placebo — Placebo matched to maralixibat will be provided as an oral solution along with 0.5-, 1.0-, and 3.0-mL sized dosing dispensers. During the double-blind dose escalation period (4 weeks), study drug will be administered once daily for 1 week and then twice daily (BID; morning and evening). During the double-blind stable dosing period (16 weeks), participants will be treated with 300 μg/kg BID or the maximum tolerated dose (determined during the double-blind dose-escalation period) of study drug. During the open-label dose escalation period (4 weeks), all participants will receive maralixibat treatment once daily for 1 week and then twice daily (BID; morning and evening). During the open-label stable dosing period (16 weeks), participants will be treated with 300 μg/kg BID or the maximum tolerated dose (determined during the open-label dose-escalation period) of maralixibat.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether the investigational treatment (maralixibat) is safe and effective in pediatric and adult participants who have cholestatic liver disease with pruritus that has been refractory to other therapies, and who have no other treatment options.

DETAILED DESCRIPTION:
This study will be conducted in multiple sites in North America, Europe, Middle East and South America.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent and assent (as applicable)
2. Age ≥6 months at time of baseline visit
3. Diagnosis of cholestatic liver disease with cholestatic pruritus based on the presence of chronic liver biochemical abnormalities (>90 days) and/or pathological evidence of progressive liver disease.
4. If taking antipruritics or ursodeoxycholic acid, the participant has to be on a stable dosing regimen (i.e., same dose and frequency in the 30 days prior to the screening visit and will continue this dosing regimen up to Week 40 [adjustment for body weight is allowed]).
5. Access to email or telephone for scheduled participant contacts and access to smart phone or tablet for PROs.
6. Ability to read and/or understand the questionnaires (both caregivers and participants ≥9 years of age).
7. For participants ≤18 years of age: Access to consistent caregiver(s) during the study.

Exclusion Criteria:

Those who meet any of the following criteria are NOT eligible to participate in the study:

1. Diagnosis of ALGS, ICP, PBC, PFIC, or PSC with native liver.
2. Active atopic dermatitis or other non- cholestatic diseases associated with pruritus that are not controlled by standard treatment and that may interfere with the severity assessment of cholestasis-associated pruritus.
3. Decompensated cirrhosis or complications of cirrhosis (e.g., esophageal or gastric variceal bleeding in the last 6 months, high-risk esophageal or gastric varices, ascites, hepatic encephalopathy, hepatorenal syndrome). Patients with compensated cirrhosis with preserved hepatic synthetic function and absence of complications are eligible.
4. Suspected or proven cholangiocarcinoma or hepatocellular carcinoma.
5. Unstable and/or serious medical disease that is likely to impair the ability to participate in all aspects of the study, confound efficacy and/or safety assessments, or result in substantially shortened life expectancy (e.g., any active malignancy including hematological malignancy, end-stage heart failure, active infection, acute and chronic diarrhea). Exceptionally, previous history of malignancy, adequately treated/in remission, that in opinion of investigator and medical monitor does not impact participant safety and participation in the study, may be allowed.
6. Laboratory results during the screening visit as follows:

   1. Platelet count ≤70,000/mm3. Patients with any condition that further increases bleeding risk are excluded.
   2. Albumin <30 g/L
   3. INR ≥1.5 (after intravenous or subcutaneous supplementation of vitamin K)
   4. Total bilirubin >10 mg/dL
   5. ALT >10× ULN
7. Use of an IBAT inhibitor within 8 weeks prior to the screening visit.
8. Known intolerance/hypersensitivity to maralixibat or its excipients.
9. History of nonadherence to medical regimens, unreliability, medical condition, mental instability, or cognitive impairment that, in the opinion of the investigator, could compromise the validity of informed consent, compromise the safety of the participant, or lead to nonadherence with the study protocol or inability to conduct the study procedures.

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-10-14 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Mean change in the ItchRO(Obs) severity score | From baseline to average of week 13 to week 20
  ItchRO(Obs) severity score = Itch Reported Outcome Observer assessment severity score; scale between 0 (not itchy at all) and 4 (extremely itchy); the lower the score the better.

SECONDARY OUTCOMES:
Mean change in total sBA (serum bile acid) level | From baseline to average of week 12 and week 20

CONTACTS AND LOCATIONS:
Locations (35):
- United States (14):
  - Children's Hospital Los Angeles (CHLA), Los Angeles, California
  - Stanford Children's Health in Palo Alto, Palo Alto, California
  - Lurie Children's Hospital, Chicago, Illinois
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - NYU Langone Health, New York, New York
  - Mount Sinai Hospital, New York, New York
  - Morgan Stanley Children's Hospital - NewYork Presbyterian, New York, New York
  - Science 37, Inc (Remote-homebase Telemedicine), Morrisville, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
- Brazil (3):
  - Hospital de Criança de Brasília (HCB), Brasília
  - Hospital da Criança Santo Antonio, Porto Alegre
  - Hospital Sírio-Libanês, São Paulo
- Stollery Children's Hospital, Edmonton, Alberta, Canada
- France (3):
  - Hôpital Femme Mère Enfant, Lyon
  - Hôpitaux Universitaires de Marseille Timone, Marseille
  - Hôpital Kremlin Bicêtre, Paris
- Germany (2):
  - Universitätsklinikum Hamburg Eppendorf - Klinik für Kinder- und Jugendmedizin, Hamburg
  - LMU Klinikum - Kinderklinik und Kinderpoliklinik im Dr. von Haunerschen Kinderspital, Munich
- Italy (3):
  - Azienda Ospedaliera Papa Giovanni XXIII, Bergamo
  - ISMETT - Istituto Mediterraneo per i Trapianti e Terapie ad Alta Specializzazione, Palermo
  - Ospedale Pediatrico Bambino Gesu, Rome
- Hotel Dieu de France, Beirut, Lebanon
- Mexico (2):
  - Hospital Infantil de México Federico Gómez, Mexico City
  - Consultario de Joshue David Covarrubias Esquer, Zapopan
- Instytut Pomnik Centrum Zdrowia Dziecka, Warsaw, Poland
- King Faisal Specialist Hospital & Research Center, Riyadh, Saudi Arabia
- Spain (3):
  - Hospital Sant Joan de Deu, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitario La Paz, Madrid
- King's College Hospital NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mirum Pharmaceuticals homepage — https://mirumpharma.com/